CLINICAL TRIAL: NCT04166747
Title: Effect of Virtual Reality Based Intervention on Functional Fitness and Quality of Life of Older Population: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality on Functional Fitness and Quality of Life of Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shabbir Syed Abdul, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N201906048
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Aging; Happiness; Quality of Life
Keywords: virtual reality; older population; functional fitness; quality of life; happiness

STUDY DESIGN:
Intervention Model Description: Intervention study with 2 parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants in this group will receive virtual reality based intervention for 15 minutes at a time, twice in a week for six weeks.
  Interventions: Other: Virtual Reality experience
- Control Group (No Intervention): The participants in this group will not receive virtual reality based intervention for six weeks.

INTERVENTIONS:
Other: Virtual Reality experience — Participants will receive virtual reality based experience and will be assessed for its influence on happiness, functional fitness components and quality of life of older age groups.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess the influence of virtual reality (VR) on the different parameters, happiness, quality of life and functional fitness, among older population. The study aims to conduct a randomized controlled trial, where the participants in intervention group will use VR and those in control group do not use VR.

DETAILED DESCRIPTION:
This study aims to conduct a randomized control trial, on 60 older age group participants, and perform the functional fitness test based on the protocol developed by Rikli and Jones, before and after the VR intervention. The functional fitness tests include evaluation of upper body strength, lower body strength, cardiorespiratory endurance, upper body flexibility test, lower body flexibility test, balance, agility test. They will be randomly assigned to the intervention group, receiving the VR program, and the control group who will not receive the VR program. The participants in the intervention group will be asked to use the VR device for 15 minutes, twice a week for 6 weeks, along with their daily routine activities. Control group will carry out the daily routine activities, without the intervention. The change in the quality of life (QOL) and happiness, for both control and intervention groups, will be assessed through EuroQol 5 dimensions 3 level questionnaire (EQ-5D-3L), mini version of Chinese happiness Inventory questionnaire, respectively, to filled at recruitment and follow-up after 6 weeks. The effect of the VR programs will be determined by the comparison of performance, for the functional fitness tests before and after the intervention and also, for the differences between the control and intervention groups

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 60 years or older and approach TMU aging center.
* Able to understand Mandarin Chinese.
* Gives informed consent to participate
* No past or current history of serious medical disease
* Ability to perform activities of daily living
* Understands the intent of the study

Exclusion Criteria:

* Participants aged below 60 years of age.
* Not able to understand Mandarin Chinese.
* Does not gives informed consent to participate
* Past or current history of serious medical disease
* Inability to perform activities of daily living
* Does not understand the intent of the study

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Quality of life | At enrollment and at 6 weeks after enrollment
  Comparison of changes in the quality of life through the questionnaire EQ-5D-3L
Measurement of functional fitness components | At enrollment and at 6 weeks after enrollment
  Comparison of changes in the muscle strength through the functional fitness tests.
Measurement of Happiness | At enrollment and at 6 weeks after enrollment
  Comparison of changes in the happiness through the questionnaire mini version of Chinese Happiness Inventory.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taipei City, Taiwan

REFERENCES:
- [Derived] Barsasella D, Liu MF, Malwade S, Galvin CJ, Dhar E, Chang CC, Li YJ, Syed-Abdul S. Effects of Virtual Reality Sessions on the Quality of Life, Happiness, and Functional Fitness among the Older People: A Randomized Controlled Trial from Taiwan. Comput Methods Programs Biomed. 2021 Mar;200:105892. doi: 10.1016/j.cmpb.2020.105892. Epub 2020 Nov 29. PMID 33280934